CLINICAL TRIAL: NCT00171821
Title: A One Year, Open-label, Single-arm, Multi-center Trial Evaluating the Efficacy and Safety of Oral ICL670 (20 mg/kg/Day) in Patients Diagnosed With Transfusion-dependent Iron Overload
Brief Title: A Study Assessing the Efficacy and Safety of Deferasirox in Patients With Transfusion-dependent Iron Overload
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2409; 2004-003953-16 (EudraCT Number); NCT00565578 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2013-06

CONDITIONS: Transfusion-dependent Iron Overload
Keywords: Thalassemia; Myelodysplastic Syndrome; MDS; Sickle cell; Diamond-Blackfan anemia; Transfusion; Anemia; Fanconi; Chelation; Deferasirox
MeSH Terms: conditions — Thalassemia; Myelodysplastic Syndromes; Anemia, Diamond-Blackfan; Anemia | interventions — Deferasirox

ARMS (1):
- ICL670 (Deferasirox) (Experimental)
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox
  Other Names: ICL670

SUMMARY:
This study uses a single arm, multi-center, open-label trial design. The study will assess the efficacy and safety of 52 weeks of treatment with deferasirox (ICL670) in patients with evidence of transfusion induced iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with transfusion-dependent anemias (independent of underlying condition) with transfusional iron overload as shown by a serum ferritin level of ≥ 1000 ng/ml
* Patients of either gender and aged ≥ 2 years
* Female patients who have reached menarche and who are sexually active must use an effective method of contraception, or must have undergone clinically documented total hysterectomy and/or ovariectomy, or tubal ligation.

Additional Inclusion Criteria for Adult Patients:

* Written informed consent by the patient

Additional Inclusion Criteria for Pediatric Patients:

* The definition of the term "pediatric" will be in accordance with local legislation. Parents or legal guardians will be fully informed by the investigator as to the requirements of the study. The pediatric patients themselves will be informed according to their capabilities in a language and terms that they are able to understand. Written informed consent will be obtained from their parents or legal guardians on the patient's behalf in accordance with the national legislation. If capable, all patients should also personally sign their written informed assent.

Exclusion Criteria:

* Non-transfusional hemosiderosis
* Patients with clinical evidence supporting the need for intensive chelation, based on the investigator's judgment
* Patients with mean levels of alanine aminotransferase (ALT) > 300 U/l
* Patients with uncontrolled systemic hypertension
* Patients with serum creatinine above the upper limit of normal (ULN)
* Significant proteinuria as indicated by a urinary protein/creatinine ratio > 0.5 (mg/mg) in second-voiding urine samples taken at both visits 1 and 2. A third sample is to be taken from patients in whom one ratio is > 0.5 (mg/mg) and one is ≤ 0.5 (mg/mg) and patients in whom the urinary protein/creatinine ratio is > 0.5 (mg/mg) in two of the three determinations are also to be excluded.
* History of nephrotic syndrome
* Patients with 3rd atrioventricular (A-V) block, clinically relevant Q-T interval prolongation as well as patients requiring treatment with digoxin and similar compounds or drugs which may induce prolongation of the Q-T interval
* Patients with a previous history of clinically relevant ocular toxicity related to iron chelation
* Systemic diseases (cardiovascular, renal, hepatic, etc.) which would prevent the patient from undergoing study treatment
* Patients with psychiatric or addictive disorders which prevent them from giving their informed consent or undergoing study treatment
* Pregnant or breast feeding patients
* Patients treated with systemic investigational drugs within the past 4 weeks or topical investigational drugs within the past 7 days
* Any other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug. The investigator should be guided by evidence of any of the following:

  * history of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding;
  * history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
  * history of pancreatic injury or pancreatitis; indications of impaired pancreatic function/injury as indicated by abnormal lipase or amylase;
  * history or presence of impaired renal function as indicated by creatinine or blood urea nitrogen (BUN) values equal or above ULN;
  * history of urinary obstruction or difficulty in voiding.
* History of non-compliance to medical regimens and patients who are considered potentially unreliable and/or not cooperative
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the run-in period
* Patients with positive test to HIV
* Life expectancy of < 1 year

Exclusion Criteria for Pediatric Patients:

* Patient body weight which prevents the use of the smallest tablet strength (i.e. 125 mg) for proper dosing

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1784 (Actual)
Dates: Start 2005-04; Primary Completion 2009-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To evaluate if fixed starting doses of ICL670, based on transfusion history and subsequent dose titration can provide clinically acceptable chelation as measured by serum ferritin | at baseline and at 52 weeks

SECONDARY OUTCOMES:
To evaluate the safety and tolerability profile of in patients treated for up to 52 weeks | Monthly
Evaluate efficacy, tolerabilty and safety in the subgroup of patients with baseline LIC < 7 mg Fe/g dw | Monthly
Evaluate the relationship between serum ferritin and potential surrogate markers | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (97):
- Australia (7):
  - Novartis Investigative Site, Adelaide
  - Novartis Investigative Site, Camperdown
  - Novartis Investigative Site, Clayton
  - Novartis Investigative Site, Melbourne
  - Novartis Investigative Site, Perth
  - Novartis Investigative Site, South Brisbane
  - Novartis Investigative Site, Westmead
- Austria (3):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (5):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Godinne
  - Novartis Investigative Site, La Louvière
  - Novartis Investigative Site, Leuven
- China (3):
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Nanjing
  - Novartis Investigative Site, Shanghai
- Denmark (4):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Hillerød
- Novartis Investigative Site, Cairo, Egypt
- France (12):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (13):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Braunschweig
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Frieburg
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Ulm
- Greece (4):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Larissa
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Hong Kong, Hong Kong
- Israel (3):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
- Italy (14):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Brindisi
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Cona
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Orbassano
  - Novartis Investigative Site, Palermo
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Reggio Calabria
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Sassari
- Novartis Investigative Site, Hazmiyeh, Lebanon
- Malaysia (2):
  - Novartis Investigative Site, Kota Bharu
  - Novartis Investigative Site, Kuala Lumpur
- Novartis Investigative Site, Nijmegen, Netherlands
- South Africa (2):
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Parktown
- Novartis Investigative Site, Seoul, South Korea
- Spain (5):
  - Novartis Investigative Site, Barakaldo
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Switzerland (2):
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Zurich
- Taiwan (2):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chaingmai
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (5):
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Sheffield

REFERENCES:
- [Derived] Porter JB, El-Alfy M, Viprakasit V, Giraudier S, Chan LL, Lai Y, El-Ali A, Han J, Cappellini MD. Utility of labile plasma iron and transferrin saturation in addition to serum ferritin as iron overload markers in different underlying anemias before and after deferasirox treatment. Eur J Haematol. 2016 Jan;96(1):19-26. doi: 10.1111/ejh.12540. Epub 2015 Jun 23. PMID 25691036
- [Derived] Lee JW, Yoon SS, Shen ZX, Ganser A, Hsu HC, El-Ali A, Habr D, Martin N, Porter JB. Hematologic responses in patients with aplastic anemia treated with deferasirox: a post hoc analysis from the EPIC study. Haematologica. 2013 Jul;98(7):1045-8. doi: 10.3324/haematol.2012.077669. Epub 2013 Apr 12. PMID 23585526
- [Derived] Pennell DJ, Porter JB, Cappellini MD, Chan LL, El-Beshlawy A, Aydinok Y, Ibrahim H, Li CK, Viprakasit V, Elalfy MS, Kattamis A, Smith G, Habr D, Domokos G, Roubert B, Taher A. Continued improvement in myocardial T2* over two years of deferasirox therapy in beta-thalassemia major patients with cardiac iron overload. Haematologica. 2011 Jan;96(1):48-54. doi: 10.3324/haematol.2010.031468. Epub 2010 Nov 11. PMID 21071497
- [Derived] Lee JW, Yoon SS, Shen ZX, Ganser A, Hsu HC, Habr D, Domokos G, Roubert B, Porter JB; EPIC study investigators. Iron chelation therapy with deferasirox in patients with aplastic anemia: a subgroup analysis of 116 patients from the EPIC trial. Blood. 2010 Oct 7;116(14):2448-54. doi: 10.1182/blood-2010-01-261289. Epub 2010 Jun 21. PMID 20566896
- [Derived] Pennell DJ, Porter JB, Cappellini MD, El-Beshlawy A, Chan LL, Aydinok Y, Elalfy MS, Sutcharitchan P, Li CK, Ibrahim H, Viprakasit V, Kattamis A, Smith G, Habr D, Domokos G, Roubert B, Taher A. Efficacy of deferasirox in reducing and preventing cardiac iron overload in beta-thalassemia. Blood. 2010 Mar 25;115(12):2364-71. doi: 10.1182/blood-2009-04-217455. Epub 2009 Dec 8. PMID 19996412
- [Derived] Cappellini MD, Porter J, El-Beshlawy A, Li CK, Seymour JF, Elalfy M, Gattermann N, Giraudier S, Lee JW, Chan LL, Lin KH, Rose C, Taher A, Thein SL, Viprakasit V, Habr D, Domokos G, Roubert B, Kattamis A; EPIC Study Investigators. Tailoring iron chelation by iron intake and serum ferritin: the prospective EPIC study of deferasirox in 1744 patients with transfusion-dependent anemias. Haematologica. 2010 Apr;95(4):557-66. doi: 10.3324/haematol.2009.014696. Epub 2009 Nov 30. PMID 19951979